CLINICAL TRIAL: NCT02839187
Title: Neuro Imaging and Multimodal Alzheimer's Disease
Acronym: NIMAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07 306 02
Record Dates: First submitted 2016-07-04; First posted 2016-07-20 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Alzheimer Disease (Experimental): Patients will have Neuroimaging by Florbetapir (AV-45)-positron emission tomography
  Interventions: Radiation: Neuroimaging
- Controls patients (Active Comparator): Controls will have neuroimaging by AV45-positron emission tomography
  Interventions: Radiation: Neuroimaging

INTERVENTIONS:
Radiation: Neuroimaging — AV45-positron emission tomography

SUMMARY:
The present study aimed at measuring cerebral changes in Alzheimer Disease (AD) patients, who responded to strict physiological criteria typical of AD pathology. The objective of the present study was to identify the earliest alterations in cerebral connections that could contribute to the initial episodic memory impairment.

ELIGIBILITY:
Inclusion Criteria:

For all subjects :

* Capacities visual, auditory (authorized devices) and oral or written expression sufficient for the proper performance of tests
* Obtain informed written consent of the subject

Patients with AD :

* Outpatient accompanied by a "helping"
* No parenchymal lesions allowing isolation explain the symptoms on brain MRI (T1 and T2) carried more than 6 months prior to enrollment in the study. Patients with more than three hyperintense white matter or visible lacunar infarction or T2 FLAIR will not be included in the study.
* probable Alzheimer's disease diagnosis par with international standards
* Illness in a mild stage (CDR 1, 24 ≥ Mini-Mental State Examination (MMSE)> 18)
* activity of daily living (ADL) 4 items> 1/4

Patients with Alzheimer's disease at a pre-dementia stage:

* Alzheimer's Diagnosis pre-dementia based on the search criteria
* Illness in a mild stage (CDR 0.5, 30 ≥ MMSE ≥ 25)
* ADL items ≤ 4 1/4

Control subjects :

* 30 ≥ MMSE ≥ 27
* perfect autonomy in daily living (IADL = 0, CDR = 0)
* Neuropsychological evaluation not highlighting of impaired cognitive performance with focus on memory performance
* No parenchymal lesions on brain MRI.
* Lack of family history (first degree) of Alzheimer's disease

Exclusion Criteria:

* Subjects with a contra-indication to MRI (carrying a pacemaker or cardiac defibrillator, implanted a material activated by an electrical, magnetic or mechanical carriers hemostatic clips intracerebral aneurysms or carotid artery , holders of orthopedic implants, claustrophobia)
* Subjects with clinically significant gastrointestinal, renal, hepatic, endocrine, or cardiovascular
* Subjects with a psychiatric disorder or progressive neurological
* French Language level insufficient to be appropriately involved in neurophysiological evaluation
* less than 5 years Education (insufficient understanding level to participate in the study)
* Administrative problems: unable to give informed about information, not covered by a social security system
* Hypersensitivity to the active substance or to any of the excipients
* unbalanced diabetes mellitus
* Subjects treated by a non-steroidal anti-inflammatory

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
fixing the AV-45 during PET | baseline
  compare fixing the AV-45 during a examination emission tomography (PET) between three different groups: healthy subjects, patients with Alzheimer's disease and a mild stage patients of Alzheimer's disease at a pre-dementia stage

SECONDARY OUTCOMES:
Deposition of amyloid protein | baseline
  Correlation between the deposition of amyloid protein assessed by metabolic imaging (AV-45) and cognitive performance in a group of patients with Alzheimer's disease compared to a control group
Standard Cognitive function | Baseline
  no memory performance: language (OD 80), executive functions (TMT A and B, evocations formal and categorical lexical, Stroop test, Pyramid-palm tree test Visual and Verbal) praxis visuo-constructive (copy of the figure of Rey) ; working memory (span of front and back numbers, subtest of the WAIS code-III)
Specific memory evaluation | Baseline
  anterograde verbal memory (test Gröber and Buschke), memory unique items (visual DMS48), semantic memory (sub-test information of theWechsler Adult Intelligence Scale (WAIS))

CONTACTS AND LOCATIONS:
Overall Officials: PARIENTE Jérémie, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nemmi F, Saint-Aubert L, Adel D, Salabert AS, Pariente J, Barbeau EJ, Payoux P, Peran P. Insight on AV-45 binding in white and grey matter from histogram analysis: a study on early Alzheimer's disease patients and healthy subjects. Eur J Nucl Med Mol Imaging. 2014 Jul;41(7):1408-18. doi: 10.1007/s00259-014-2728-4. Epub 2014 Feb 27. PMID 24573658
- [Result] Saint-Aubert L, Nemmi F, Peran P, Barbeau EJ, Payoux P, Chollet F, Pariente J. Comparison between PET template-based method and MRI-based method for cortical quantification of florbetapir (AV-45) uptake in vivo. Eur J Nucl Med Mol Imaging. 2014 May;41(5):836-43. doi: 10.1007/s00259-013-2656-8. Epub 2013 Dec 19. PMID 24435769
- [Result] Saint-Aubert L, Barbeau EJ, Peran P, Nemmi F, Vervueren C, Mirabel H, Payoux P, Hitzel A, Bonneville F, Gramada R, Tafani M, Vincent C, Puel M, Dechaumont S, Chollet F, Pariente J. Cortical florbetapir-PET amyloid load in prodromal Alzheimer's disease patients. EJNMMI Res. 2013 Jun 3;3(1):43. doi: 10.1186/2191-219X-3-43. PMID 23731789